CLINICAL TRIAL: NCT05795985
Title: Role of Faecal Calprotectin in Patients Presenting to the Emergency Department With Abdominal Pain
Brief Title: Role of Faecal Calprotectin in Patients With Abdominal Pain
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, OJETTI VERONICA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4183
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- abdominal pain: patients with abdominal pain
  Interventions: Diagnostic Test: calprotectin levels

INTERVENTIONS:
Diagnostic Test: calprotectin levels — dosage of calprotectin levels in patients with abdominal pain

SUMMARY:
The evaluation of patients with abdominal pain is a challenge for the emergency physician and the selection of patients for second-level radiological examinations or endoscopic procedures is not always easy to perform. Faecal calprotectin could be a useful diagnostic marker to distinguish between "organic" or "functional" form and its determination could be helpful to select patients for further examinations, in the context of emergency setting.

ELIGIBILITY:
Inclusion Criteria:

* patients with abdominal pain and/or diarrhea and/or rectal bleeding

Exclusion Criteria:

* patients with age < 18 years
* pregnant women;
* patients with oncological, cardiological, nephrological terminal diseases;
* patients on antibiotic therapy or who have taken it during the last month;
* patients with a history of colic resection or gastrointestinal surgery;
* patients with a previous diagnosis of inflammatory bowel disease (Crohn's disease, ulcerative colitis)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with abdominal pain and/or diarrhea and/or rectal bleeding accessing the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
inflammation | 3 days
  assess the degree of intestinal inflammation by fecal calprotectin assay in patients with abdominal pain

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy